CLINICAL TRIAL: NCT03146975
Title: Effects of Non-surgical Periodontal Treatment on Gingival Beta Defensins in Different Clinical Conditions : a Short-term Clinica Trial
Brief Title: Effects of Gum Disease Treatment on Host Defense Factors
Acronym: PETREBED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Fernando O Costa, Head of periodontology, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beta defensins in periodontics
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Periodontitis; Diabetes Mellitus
Keywords: Beta-defensins; Chronic periodontitis; Diabetes mellitus; Non-surgical periodontal therapy
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy (No Intervention)
- Periodontitis without diabetes (Experimental)
  Interventions: Procedure: Non-surgical periodontal treatment
- Periodontitis compensated diabetes (Experimental)
  Interventions: Procedure: Non-surgical periodontal treatment
- Periodontitis decompensated diabetes (Experimental)
  Interventions: Procedure: Non-surgical periodontal treatment
- Compensated diabetes non periodontitis (No Intervention)
- Decompensated diabetes non periodontitis (No Intervention)

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Quadrant-wise ultrasonic debridement followed by manual scaling and root planing under local anesthesia provided in weekly sections. Oral hygiene instructions.
  Arms: Periodontitis compensated diabetes; Periodontitis decompensated diabetes; Periodontitis without diabetes

SUMMARY:
Human immune system produces many different factors, which will influence health-disease statuses. This partially explains why under similar conditions only some people become sick. Therefore, specific analyses of such factors in healthy and diseased patients are crucial for a better knowledge about diseases development and successful treatments. Human beta defensins (hBD) may have a key role in patient's susceptibility to gum diseases. In the lab, high levels of sugar (glucose) could inhibit their expression and contribute to the occurrence of infections associated with diabetic wounds. This study will evaluate if treatment of the most common gum disease in adults influences production of beta defensins by gingiva. Also, clinical improvements and treatment effects on blood glycemic levels will be monitored throughout a 2-month period. Patients with or without gum diseases and with or without diabetes mellitus will be able to participate. After a complete oral examination to determine periodontal status, gingival fluid samples will be collected using paper strips. These samples will be collected before and also two-months after oral treatment and will be analyzed by an immune-enzymatic test named ELISA (Enzyme-Linked Immunosorbent Assay). In weekly sections, one trained specialist will performed treatment of gum diseases under local anesthesia using hand-instruments. Researchers hypothesized that a) levels of defensins would be lower in the presence of periodontal disease when compared to a healthy periodontal condition; b) diabetes would influence production of these immune protective factors; and c) treatment would provide a greater beneficial amount of defensins.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally healthy individuals: at least 15 natural teeth, periodontal pocket depth (PPD) ≤ 3mm e absence of bleeding on probing.
* Periodontitis individuals: at least 15 natural teeth and at least 4 teeth with one or more periodontal sites showing combined PPD ≥ 4mm and clinical attachment level (CAL) ≥ 3mm.
* Compensated diabetic individuals: compensated type 2 diabetes mellitus
* Decompensated diabetic individuals: decompensated type 2 diabetes mellitus (glycated hemoglobin HbA1c >7%)

Exclusion Criteria:

* Past or actual systemic diseases other than diabetes type 2 in the diabetic groups
* Gingivitis
* Gingival overgrowth
* Necrotizing periodontal diseases
* Pregnant or lactating
* smokers or former-smokers
* medication that can influence periodontal status or host response to periodontal therapy
* periodontal therapy in the past 6 months from baseline
* use of systemic or local antibiotics or anti-inflammatory drugs within 3 months prior baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03-02 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Changes in beta defensins 1, 2 and 3 | Baseline and 60 days
  Increase in the expression of beta defensins 1, 2 and 3 in gingival crevicular fluid samples

SECONDARY OUTCOMES:
Changes in periodontal pocket depth | Baseline and 60 days
  Reduction in mean periodontal pocket depth
Changes in blood glycemic levels | Baseline and 60 days
  Reduction in blood glucose levels and levels of glycated hemoglobin
Changes in percentage of diseased sites | Baseline and 60 days
  Reduction in the percentage of sites showing PPD>4mm and/or bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Fernando O Costa, PhD, Principal Investigator — Dean periodontics department
Locations (1):
- Federal university of minas gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only data without identification will be submitted to statistical analysis.